CLINICAL TRIAL: NCT05393544
Title: Digitally Assisted Virtual Recovery Coach to Improve Inpatient Alcohol Withdrawal Management: A Proof-of-concept Pilot Study
Brief Title: Digitally Assisted Recovery Coach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Director, Division of Addiction Psychiatry, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000731
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Alcohol Use Disorder; Alcohol Withdrawal
Keywords: alcohol use disorder; peer recovery coach; smartphone app
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention utilizes an existing care coordination smartphone app to allow participants to engage with a recovery coach during and after an inpatient admission to an inpatient withdrawal management facility (i.e. detox).
  Interventions: Behavioral: Digitally assisted peer recovery coach

INTERVENTIONS:
Behavioral: Digitally assisted peer recovery coach — The certified peer recovery coach utilized an existing care coordination smartphone app to provide support to the patient during and after an inpatient detoxification treatment for alcohol use disorder. The coach utilized the telephone or text messages to send daily motivational messages, remind about upcoming appointments, and checked-in if responses were concerning. Follow-up by the coach continued for 30 days.

SUMMARY:
The aims of this proof-of-concept study are to determine the feasibility of 1) using a smartphone app ("Lifeguard") to facilitate engagement with a peer recovery coach, 2) monitoring post-detox using a modified Brief Addiction Monitor, and 3) assessing linkage to care post-detox.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65
* Diagnosis of DSM-5 alcohol use disorder
* Admitted to Brigham and Women's Faulkner Hospital (BWF) inpatient Addiction Recovery Program to treat alcohol withdrawal
* Own either an iOS or Android smartphone device
* Have an active email address
* English speaking

Exclusion Criteria:

* Inability to provide informed consent due to delirium or other cognitive impairments
* Current psychosis, suicidality or homicidality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of coach engagement | 30 days
  The proportion and the number of days of participants engaging with the coach during and after detoxification.

SECONDARY OUTCOMES:
Feasibility of monitoring clinical status | 30 days
  The proportion and the number of days of participants responding to prompts during and after detoxification.
Linkage to care | 30 days
  The proportion of participants successfully linking to care after discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Faulkner Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suzuki J, Loguidice F, Prostko S, Szpak V, Sharma S, Vercollone L, Garner C, Ahern D. Digitally Assisted Peer Recovery Coach to Facilitate Linkage to Outpatient Treatment Following Inpatient Alcohol Withdrawal Treatment: Proof-of-Concept Pilot Study. JMIR Form Res. 2023 Jul 5;7:e43304. doi: 10.2196/43304. PMID 37405844